CLINICAL TRIAL: NCT02324972
Title: The KINSHIP Trial: A Randomized, Double-Blind, Multicenter, Placebo-Controlled Phase 2 Study to Evaluate the Efficacy and Safety of AQX-1125 in Subjects With Atopic Dermatitis by Targeting the SHIP1 Pathway
Brief Title: Pilot Efficacy and Safety Study of AQX-1125 in Atopic Dermatitis
Acronym: KINSHIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aquinox Pharmaceuticals (Canada) Inc. (Industry)
Collaborators: Innovaderm Research Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AQX-1125-204
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Results first posted 2018-10-05 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2017-12

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Eczema; AD; AQX-1125; SHIP1
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — 4-(4-(aminomethyl)-7a-methyl-1-methylideneoctahydro-1H-inden-5-yl)-3-(hydroxymethyl)-4-methylcyclohexan-1-ol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AQX-1125 (Experimental): 1 x AQX-1125 Capsule daily
  Interventions: Drug: AQX-1125
- Placebo (Placebo Comparator): 1 x placebo capsule daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AQX-1125 — Synthetic SHIP1 activator
  Arms: AQX-1125
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the effect of 12 weeks of treatment with once daily administration of AQX-1125 compared to placebo on change from baseline in Total Lesion Symptom Score in subjects with mild to moderate atopic dermatitis

DETAILED DESCRIPTION:
One of the causative factors for the inflammatory response observed in AD is the release of chemokines and other chemoattractant factors followed by recruitment of inflammatory cell subtypes (10). IL-16, a Langerhans cells (LC)-derived chemoattractant cytokine for CD4+ cells, RANTES, monocyte chemotactic protein (MCP-4) and eotaxin are overexpressed in epidermal keratinocytes from AD subjects and may contribute to the chemotaxis of eosinophils, macrophages and Th2-lymphocytes (11).

Since the activation of SHIP1 by AQX-1125 results in the inhibition of inflammatory cell chemotaxis and reduction of pro-inflammatory cytokine synthesis, this study hypothesized that AQX-1125 would improve AD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged from 18 to 65 years old
2. Confirmed clinical diagnosis of active atopic dermatitis (AD) according to the Hanifin and Rajka criteria
3. At least a 6 months history of atopic dermatitis.
4. Body Surface Area (BSA) covered with atopic dermatitis of 1% or more
5. Mild or moderate atopic dermatitis (IGA score of 2 or 3).
6. TLSS of 5 or more at Day 0.
7. Subject must use a non-medicated emollient daily for at least (≥) 7 days prior to Day 0 and should continue using that same emollient, at the same frequency, throughout the study.

Exclusion Criteria:

1. Female subject who is pregnant or breast-feeding
2. Unstable or clinically infected atopic dermatitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Wang, MD, Study Director — Aquinox Pharamceuticals Inc
Locations (1):
- AQX-Innovaderm site, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 1 x placebo capsule daily
  Placebo: Double blind placebo capsule
Period: Overall Study
Arm/Group | AQX-1125 | Placebo
Started | 26 | 28
Completed | 19 | 23
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Placebo: 1 x placebo capsule daily
  Placebo
- Total: Total of all reporting groups
Arm/Group | AQX-1125 | Placebo | Total
Number analyzed (Participants) | 26 | 28 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 28 | 54
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 14 | 32
  Male | 8 | 14 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 24 | 28 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 19 | 25 | 44
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 26 | 28 | 54
Weight [Mean (Standard Deviation); unit: kg] | 72.96 (19.44) | 76.30 (16.06) | 74.69 (17.67)
BMI [Mean (Standard Deviation); unit: kg/m2] | 26.4 (6.17) | 27.1 (5.28) | 26.8 (5.68)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Lesion Symptom Score (TLSS)
Description: The TLSS is an assessment of the severity of each of the following three signs: erythema, papulation/infiltration, excoriation and lichenification. Each of these items are rated using a 4-point scale severity where 0 is clear, 1 = mild, 2= moderate and 3 = severe. These ratings are then added to create a total score ranging from 0 to 12
Time Frame: 12 weeks
Population: The intent to treat analysis population (ITT) is the set of subjects who were randomized and received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AQX-1125 | Placebo
Number analyzed (Participants) | 26 | 28
units on a scale
  Baseline | 6.3 (1.16) | 6.6 (1.31)
  Week 12 (Change from baseline): number analyzed (Participants) | 20 | 24
  Week 12 (Change from baseline) | -1.9 (2.19) | -1.9 (2.41)
Statistical Analysis 1: Comparison: AQX-1125 vs Placebo; A sample size of 20 subjects per group was assumed to have 80% power to allow detection of a statistically significant difference in change from baseline in TLSS between the 2 groups, if the effect size was approximately less than or equal to 0.9. This is equivalent to detecting a difference of -4.5 between the 2 groups with a common standard deviation of 5. The primary analysis was doing using last observation carried forward (LOCF) imputed data; Test type: Superiority or Other; p = 0.636, ANCOVA; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-1.30 to 1.25]

2. Secondary Outcome: Change From Baseline in Investigator's Global Assessment (IGA)
Description: The IGA is a global assessment of the current state of the disease. It is a 5-point morphological assessment of overall disease severity and will be determined according to the following categories: 0 (clear), 1 (almost clear), 2 (mild), 3 (moderate) and 4 (severe).
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AQX-1125 | Placebo
Number analyzed (Participants) | 26 | 28
units on a scale
  Baseline | 2.6 (0.50) | 2.8 (0.52)
  Week 12 (Change from baseline): number analyzed (Participants) | 20 | 24
  Week 12 (Change from baseline) | -0.7 (0.98) | -0.8 (0.87)
Statistical Analysis 1: Comparison: AQX-1125 vs Placebo; Test type: Superiority or Other; p = 0.677, ANOVA; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.44 to 0.68]

3. Secondary Outcome: Change From Baseline in Eczema Area and Severity Index (EASI) Score
Description: The Eczema Area and Severity Index (EASI) quantifies the severity of a subject's atopic dermatitis based on both lesion severity and the percentage of body surface area (BSA) affected. Lesions are assessed on four domains; 1) erythema, 2) induration/papulation, 3) excoriation and 4) lichenification. Each domain is scored separately over four body regions (head/neck, upper limbs, trunk and lower limbs) on a scale of 0-3 (0 = none, 1 = mild, 2 = moderate and 3 = severe) with adjustment for the percentage of BSA involved for each body region and for the proportion of the body region relative to the whole body. The sum of these scores provides the EASI total score, ranging from 0 to 72 with a higher score indicating greater severity of atopic dermatitis.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AQX-1125 | Placebo
Number analyzed (Participants) | 26 | 28
units on a scale
  Baseline | 5.58 (3.34) | 5.35 (2.24)
  Week 12 (Change from baseline): number analyzed (Participants) | 20 | 24
  Week 12 (Change from baseline) | -2.84 (1.55) | -2.12 (3.19)
Statistical Analysis 1: Comparison: AQX-1125 vs Placebo; Test type: Superiority or Other; p = 0.802, ANOVA; Mean Difference (Final Values) = -0.219, 95% CI 2-sided [-1.983 to 1.544]

4. Secondary Outcome: Change From Baseline in Scoring Atopic Dermatitis (SCORAD) Score
Description: The severity scoring of atopic dermatitis (SCORAD) index is a standard tool to assess the atopic dermatitis (AD) severity in clinical studies. Six items; erythema, edema/papulation, oozing/crusts, excoriation, lichenification and dryness are measured on a scale from 0-3 for a total of 18 points, with a higher score indicating greater severity. The percentage of BSA affected by AD is evaluated (percentage divided by 5) and added to the total SCORAD score. Loss of sleep and pruritus are also evaluated by subjects on a visual analog scale (scores ranging from 0-10) with a higher score indicating greater severity. The sum of these measures represents the SCORAD which ranges from 0 (absent disease) to 103 (severe disease).
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AQX-1125 | Placebo
Number analyzed (Participants) | 26 | 28
units on a scale
  Baseline | 36.19 (8.70) | 37.21 (6.38)
  Week 12 (Change from baseline): number analyzed (Participants) | 19 | 24
  Week 12 (Change from baseline) | -12.06 (11.15) | -11.54 (11.49)
Statistical Analysis 1: Comparison: AQX-1125 vs Placebo; Test type: Superiority or Other; p = 0.976, ANOVA; Mean Difference (Final Values) = 0.108, 95% CI 2-sided [-7.076 to 7.292]

5. Secondary Outcome: Change From Baseline in Patient Oriented Eczema Measure (POEM) Score
Description: The POEM is a 7-item self-assessment questionnaire that assesses disease symptoms (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) on a scale ranging from 0-4 (0 = no days, 1 = 1-2 days, 2 = 3-4 days, 3 = 5-6 days, 4 = everyday). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (severe disease). High scores are indicative of more severe disease and poor quality of life.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AQX-1125 | Placebo
Number analyzed (Participants) | 26 | 28
units on a scale
  Baseline | 16.7 (6.98) | 15.9 (5.48)
  Week 12 (Change from baseline): number analyzed (Participants) | 20 | 24
  Week 12 (Change from baseline) | -5.6 (9.70) | -6.5 (5.82)
Statistical Analysis 1: Comparison: AQX-1125 vs Placebo; Test type: Superiority or Other; p = 0.233, ANOVA; Mean Difference (Final Values) = 2.52, 95% CI 2-sided [-1.68 to 6.72]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Day 0 after 1st dose of study drug until discharge from study at Week 16
Description: Adverse events were documented by the investigator as reported by the subject, and through the asking of nonleading questions by the investigator. In addition clinically significant abnormal findings from safety assessments including; vital signs, physical exam, ECG, clinical labs and ophthalmology exam were also documented as adverse events.
Arm/Group | AQX-1125 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/28
Other Adverse Events (participants affected / at risk) | 17/26 | 14/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AQX-1125 (N=26) | Placebo (N=28)
Nausea (Gastrointestinal disorders) | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Nasopharyngitis (Infections and infestations) | 6 | 6
Folliculitis (Infections and infestations) | 0 | 3
Headache (Nervous system disorders) | 7 | 4
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 4 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators shall not publish any articles or make any presentations or communications (including any written, oral, or electronic manuscript, abstract, presentation, or other publication) relating to the Services, Sponsor Information, Study Drug or other Material, Deliverables or other Developments, in whole or in part, without the prior written consent of Sponsor.